CLINICAL TRIAL: NCT04686851
Title: Predictive Value of Geriatric Oncology Screening and Geriatric Assessment in Older Patients With Solid Cancers (PROGNOSIS-RCT)
Brief Title: Predictive Value of Geriatric Oncology Screening and Geriatric Assessment in Older Patients With Solid Cancers
Acronym: PROGNOSIS-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Danish Cancer Society (Other); Academy of Geriatric Cancer (Unknown); Odense Patient Data Explorative Network (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ann-Kristine Weber Giger, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROGNOSIS-RCT; R247-A14382 (Other Grant/Funding Number: Danish Cancer Society); 20/ 17768 (Other: Region of Southern Denmark)
Record Dates: First submitted 2020-10-26; First posted 2020-12-29 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Frailty; Cancer; Age
Keywords: Frailty; Aged; Neoplasms; Cancer Patients; Geriatric Screening; Geriatric 8; Geriatric Assessment; Randomized Clinical Trial
MeSH Terms: conditions — Frailty; Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with 2 randomized 1:1 parallel study groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Comprehensive Geriatric Assessment and follow-up as add on to standard oncologic care
  Interventions: Other: Comprehensive Geriatric Assessment and follow-up
- Control (No Intervention): standard oncologic care according to national guidelines

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment and follow-up — All patients will receive standardized oncological treatment according to national guidelines. For patients randomized to the intervention arm, a full Comprehensive Geriatric Assessment (CGA) and corresponding interventions on identified health issues will be performed alongside oncologic treatment. The domains are assessed using validated tests based on a Danish version of the Geriatric Core Dataset (G-CODE). The domains are cognition, mood, comorbidity, functional status, physical status, polypharmacy, nutrition, fall risc and social support. The CGA will be performed by the PhD-student (geriatric resident) or a geriatrician together with geriatric nurses at the Department of Geriatric Medicine, OUH. Nutritional status and interventions are assessed by a dietician. A physical therapist will evaluate the physical performance as part of the CGA.
  Follow-up on initial treatment plan is scheduled to one month after baseline CGA.
  Arms: Intervention

SUMMARY:
A Randomized Clinical Trial examining the effects of Comprehensive Geriatric Assessment as an add on to oncologic treatment. Participants included are cancer patients found eligible for oncologic treatment, age 70 or more, and screened frail with the Geriatric 8 screening tool.

DETAILED DESCRIPTION:
This study aims to examine the effects of Comprehensive Geriatric Assessment and interventions on prognosis in the older frail cancer patient in a Randomized Clinical Trial design.

Patients screened frail with the Geriatric 8 screening tool, aged 70 or more, and found eligible for oncologic treatment, will be included. We plan to enrol a total of 322 cancer patients for 12 months. Participants will be allocated randomly to either interventional or control group.

Participants in the interventional group will be offered a Comprehensive Geriatric Assessment and intervention at the start-up of cancer treatment. The Comprehensive Geriatric Assessment will be an add on to standardized cancer treatment offered at the Oncologic Outpatient Clinic at Odense University Hospital.

Comprehensive Geriatric Assessment will be performed by a team consisting of a doctor, nurse and physiotherapist. If needed, referral to a dietician or an occupational therapist for further evaluation will be made. The health issues are assessed using validated tests based on a Danish version of the Geriatric Core Dataset (G-CODE). Follow-up on Comprehensive Geriatric Assessment is scheduled for one month after initial evaluation.

The randomized groups will be compared with respect to primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Living in the region of Southern Denmark
* Newly diagnosed solid tumours assessed eligible for antineoplastic treatment
* Vulnerable or frail (G8 ≤ 14)

Exclusion Criteria:

* Inability to speak or understand Danish
* Inability to give informed consent
* Already consulting geriatric outpatient clinic
* Already receiving active treatment for other coexisting solid tumours, haematologic cancers, or non-melanoma skin cancer or has received oncologic treatment the past year

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
physical function for patients receiving palliative oncologic treatment | 3 months
  measured by 30 seconds Chair Stand Test, number of repetitions in a 30 seconds time period.
unplanned hospital admissions for patients receiving adjuvant oncologic treatment | 6 months
  number of unplanned hospitalisations including admissions to Oncologic Department, Emergency Department and Medical Departments. Data will be retrieved trough review of electronic medical records.

SECONDARY OUTCOMES:
Physical functional for patients receiving curative oncologic treatment | 3 months
  measured by 30 seconds Chair Stand Test, number of repetitions in a 30 seconds time period.
Physical functional for patients receiving curative oncologic treatment | 6 months
  measured by 30 seconds Chair Stand Test, number of repetitions in a 30 seconds time period.
Physical functional for patients receiving palliative oncologic treatment | 6 months
  measured by 30 seconds Chair Stand Test, number of repetitions in a 30 seconds time period.
number of unplanned hospital admissions for patients receiving palliative oncologic treatment | 6 months
  Number of unplanned hospitalisations including admissions to Oncologic Department, Emergency Department and Medical Departments. Data will be retrieved trough review of electronic medical records.
Health-related Quality of life | 12 months
  Measured by EORTC-QLQ-C30
Health-related Quality of life | 12 months follow-up
  Measured by EORTC-QLQ-ELD14
Elderly Functional Index Score (ELFI-score) | 6 months
  Self reported functioning score. It is a composite score derived from the three scales "physical functioning", "Role functioning" and Social Functioning", from the quality of life questionnaire EORTC-QLQ-C30 and the scale "Mobility" from the quality of life questionnaire EORTC-QLQ-ELD-14. The range is (12-48), with a higher score being a better outcome.
Number of patients who experience oncologic treatment toxicity | 6 months
  Treatment toxicity grade 3+ evaluated with Common Terminology Criteria for Adverse Events
Number of patients with adherence to initial oncologic treatment plan | 6 months
  Registration of dose reductions, discontinuations and delays of intended cancer treatment.
Degree of Polypharmacy (PP) | 3 months
  Degree of polypharmacy. Polypharmacy is defined as daily use of more than 5 prescription drugs.
Number of potential Inappropriate Medications (PIM) | 3 months
  Using the Screening Tool for Older Persons Prescriptions (STOPP) criteria. Number of PIM will be registered for each patient
Number of Potential Drug Interactions (PDI) | 3 months
  Using Stockley's Drug Interaction Database. Number of PDI will be registered for each patient
Overall survival | 12 months
  Measured from Geriatric 8 screening to time of death
Cancer specific survival | 12 months
  Measured from Geriatric 8 screening to time of death in patients with residual cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Kristine W Giger, MD, Principal Investigator — Department of Geriatric Medicine, Odense University Hospital, Odense; Cecilia M Lund, MD, PhD, Study Chair — Department of Medicine, Herlev and Gentofte University Hospital, Copenhagen; Per Pfeiffer, MD, PhD, Study Chair — Department of Clinical Oncology, Odense University Hospital, Odense; Trine L Jørgensen, MD, PhD, Study Chair — Department of Clinical Oncology, Odense University Hospital, Odense; Marianne Ewertz, MD, DMSc, Study Chair — Institute of Clinical Research, University of Southern Denmark, Odense; Henrik Ditzel, MD, DMSc, Study Chair — Department og Geriatric Medicine, Odense University Hospital, Odense; Jesper Ryg, MD, PhD, Study Director — Department of Geriatric Medicine, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giger AW, Ditzel HM, Ditzel HJ, Ewertz M, Jorgensen TL, Pfeiffer P, Lund CM, Ryg J. Effects of comprehensive geriatric assessment-guided interventions on physical performance and quality of life in older patients with advanced cancer: A randomized controlled trial (PROGNOSIS-RCT). J Geriatr Oncol. 2024 Jan;15(1):101658. doi: 10.1016/j.jgo.2023.101658. Epub 2023 Nov 6. PMID 37939628
- [Derived] Giger AW, Ditzel HM, Jorgensen TL, Ditzel HJ, Mohammadnejad A, Ewertz M, Pfeiffer P, Lund CM, Ryg J. Predictive value of geriatric oncology screening and geriatric assessment of older patients with cancer: A randomized clinical trial protocol (PROGNOSIS-RCT). J Geriatr Oncol. 2022 Jan;13(1):116-123. doi: 10.1016/j.jgo.2021.07.005. Epub 2021 Aug 4. PMID 34362713